CLINICAL TRIAL: NCT01935349
Title: Evaluation of Quality of Care - Patient Empowerment Programme, HA
Acronym: QoC PEP
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Clinical Professor, The University of Hong Kong
Other Study IDs: HKCTR-1187
Record Dates: First submitted 2013-08-28; First posted 2013-09-05 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: Diabetes mellitus (DM); hypertension (HT); Hong Kong
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diabetes mellitus (DM) and hypertension (HT): Diabetes mellitus (DM) and/or hypertension (HT) patients in Hong Kong

SUMMARY:
Diabetes mellitus (DM) and hypertension (HT) are major causes of morbidity and among the top 10 causes of deaths in Hong Kong in 2008 (Department of Health 2009). The Hospital Authority (HA) has initiated service improvement through introducing the patient empowerment programme (PEP) to improve the quality of care (QOC) for DM and HT patients. The evaluation on the QOC is an essential part of the programme in order to inform future policy. The Family Medicine Unit (FMU) of the University of Hong Kong (HKU) has been appointed by the HA to carry out the evaluation of the QOC of the programme.

The Action Learning and Audit Spiral methodologies to measure whether the target standard of care intended by the PEP programme is achieved. Each PEP participating clinic and non-government organization (NGO) will be invited to complete a structured evaluation questionnaire. The data of all patients who have enrolled into the PEP for more than one year will be included in the evaluation on the process and outcomes of care. A hundred and thirty participants will be followed up by telephone to evaluate the effect of the programme in quality of life (QOL), patient enablement, and global rating of change in health condition at baseline and 6 months after enrolment. Data on the process of care will be retrieved from the HA medical records. Main Outcome Measures: The primary outcomes are the proportion of participants who have received the planned process of care and achieved the target HbA1c and blood pressure levels.

Data Analysis: Descriptive statistics on proportions meeting the QOC criteria will be calculated. The changes in clinical, service, and patient reported outcomes at 6 and 12 months will assessed by paired sample t-test. The audit cycle will be repeated annually over a period of 5 years.

Results: The QOC of the PEP programme will be determined. Areas of deficiency and possible areas for quality enhancement will be identified. Conclusion: The results of this study will provide empirical evidence on whether the HA's PEP programme can enhance QOC for patients with diabetes mellitus (DM) or hypertension (HT). The information will be used to guide service planning and policy decision making.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients who are ambulatory, have stable mental and emotional conditions, and follow up at general outpatients clinics (GOPC) and family medicine specialist clinics (FMSC) regularly will be recruited for the PEP programme.

Exclusion Criteria:

* Patients will be excluded if they have severe heart failure, end stage renal failure (ESRF) or advanced eye diseases, are unable to understand or communicate in Chinese language, or refuse to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients who have been enrolled into the PEP programme will be included in the evaluation on process of care; whereas all enrolled subjects who have been recruited for more than 12 months in the programme will be included in the evaluation on the clinical outcomes of care. An equal number of a random sample of eligible subjects who refused to take part in the PEP will be used as controls for the evaluation on the clinical outcomes of care.
Sampling Method: Probability Sample
Enrollment: 2496 (Actual)
Dates: Start 2010-09; Primary Completion 2016-09 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The proportion of clinics/NGO that have satisfied each of the set structure criteria. | Five years
  Interim analysis will evaluate the period from August, 2009 to December, 2010; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.
The proportion of patients who have complied with the criterion process of care. | Five years
  Interim analysis will evaluate the period from August, 2009 to June, 2011; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.
The proportion of DM patients who have achieved a HbA1c level <7%. | Five years
  Interim analysis will evaluate the period from August, 2009 to June, 2011; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.
The proportion of HT/ DM patients who have achieved the target blood pressure. | Five years
  Interim analysis will evaluate the period from August, 2009 to June, 2011; to December, 2011; to December, 2012; to December, 2013. Final analysis will evaluate the period from August, 2009 to December, 2014.

SECONDARY OUTCOMES:
Clinical outcomes including LDL, BMI, and cardiovascular complications. | Five years
  Baseline and 12 months for each subject; the audit cycle will be repeated annually over a period of 5 years.
Patient reported outcomes (PRO) measured by the change in SF-12v2 scores, the Patient Enablement Index (PEI) and Global Rating of Change Score (GRS) at 6 months, and change in patient's knowledge on disease at 12 months. | Five years
  Baseline and 6-month/12-month/24-month/36-month after the first administration of questionnaire.
GOPC consultation, SOPC, A&E and hospital attendance rates in the past 12 months. | Five years
  Baseline and 12 months for each subject; the audit cycle will be repeated annually over a period of 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, MD, Study Chair — Department of Family Medicine and Primary Care, Faculty of Medicine, The University of Hong Kong; William C.W. Wong, MD, Principal Investigator — Department of Family Medicine and Primary Care, Faculty of Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong Island, Hong Kong

REFERENCES:
- [Result] Wong CK, Wong WC, Lam CL, Wan YF, Wong WH, Chung KL, Dai D, Tsui EL, Fong DY. Effects of Patient Empowerment Programme (PEP) on clinical outcomes and health service utilization in type 2 diabetes mellitus in primary care: an observational matched cohort study. PLoS One. 2014 May 1;9(5):e95328. doi: 10.1371/journal.pone.0095328. eCollection 2014. PMID 24788804
- [Result] Wong CK, Wong WC, Wan YF, Chan AK, Chung KL, Chan FW, Lam CL. Patient Empowerment Programme in primary care reduced all-cause mortality and cardiovascular diseases in patients with type 2 diabetes mellitus: a population-based propensity-matched cohort study. Diabetes Obes Metab. 2015 Feb;17(2):128-35. doi: 10.1111/dom.12397. Epub 2014 Oct 20. PMID 25251664
- [Result] Wong CK, Wong WC, Wan YF, Chan AK, Chan FW, Lam CL. Patient Empowerment Programme (PEP) and Risk of Microvascular Diseases Among Patients With Type 2 Diabetes in Primary Care: A Population-Based Propensity-Matched Cohort Study. Diabetes Care. 2015 Aug;38(8):e116-7. doi: 10.2337/dc14-2213. No abstract available. PMID 26207061
- [Result] Wong CK, Wong WC, Wan EY, Wong WH, Chan FW, Lam CL. Increased number of structured diabetes education attendance was not associated with the improvement in patient-reported health-related quality of life: results from Patient Empowerment Programme (PEP). Health Qual Life Outcomes. 2015 Aug 12;13:126. doi: 10.1186/s12955-015-0324-3. PMID 26264130
- [Result] Wong CK, Wong WC, Wan EY, Chan AK, Chan FW, Lam CL. Macrovascular and microvascular disease in obese patients with type 2 diabetes attending structured diabetes education program: a population-based propensity-matched cohort analysis of Patient Empowerment Programme (PEP). Endocrine. 2016 Aug;53(2):412-22. doi: 10.1007/s12020-015-0843-z. Epub 2016 Jan 19. PMID 26785847
- [Result] Wong CK, Wong WC, Wan YF, Chan AK, Chan FW, Lam CL. Effect of a structured diabetes education programme in primary care on hospitalizations and emergency department visits among people with Type 2 diabetes mellitus: results from the Patient Empowerment Programme. Diabet Med. 2016 Oct;33(10):1427-36. doi: 10.1111/dme.12969. Epub 2015 Oct 27. PMID 26433212
- [Result] Wong CK, Lam CL, Wan EY, Chan AK, Pak CH, Chan FW, Wong WC. Evaluation of patient-reported outcomes data in structured diabetes education intervention: 2-year follow-up data of patient empowerment programme. Endocrine. 2016 Nov;54(2):422-432. doi: 10.1007/s12020-016-1015-5. Epub 2016 Sep 13. PMID 27623970